CLINICAL TRIAL: NCT00800189
Title: A Prospective Evaluation of the Informational Content of Setup Verification Images for Patients Receiving Breast Radiation Therapy Tangentially With or Without Supraclavicular Treatment
Brief Title: Evaluation of the Informational Content of Setup Verification Images for Patients Receiving Breast Radiation Therapy (Anterior EPI)
Acronym: Anterior EPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Elaine Wai, BCCA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BCCA002
Record Dates: First submitted 2008-11-28; First posted 2008-12-02 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Anterior electronic portal images (EPI) — EPI's are taken for the first three consecutive days of treatment to detect set-up errors.

SUMMARY:
The purpose of this study is to determine if an alternative imaging protocol done at the time of radiotherapy treatments for patients with breast cancer can improve accuracy in patient set-up.

DETAILED DESCRIPTION:
Accurate patient positioning is critical in Radiation Therapy. Electronic imaging is used to compare a patient's actual treatment position, with that which was planned from an initial CT scan. Radiation Therapists compare planned and actual images using analysis software to determine if differences are within acceptable tolerances. At the VIC, we use 3 different breast imaging protocols depending on the patient set-up and treatment technique. Findings from our recent retrospective planning study show that our current electronic imaging protocols miss some clinically significant patient set-up errors, particularly in the medial/lateral direction, and that these errors can be better detected with the use of an anterior image. The purpose of this study is to test these findings prospectively in clinical practice, through the direct comparison of our current protocols with a proposed new protocol, which would include an anterior electronic portal image (EPI).

ELIGIBILITY:
Inclusion Criteria:

* All patients (male or female) receiving tangential breast/chest wall radiotherapy only, or three or four field breast/chest wall and nodal radiotherapy will be eligible.

Exclusion Criteria:

* Those patients receiving partial breast treatment, those patients requiring an electron match field, those on another breast cancer radiotherapy trial, those who require radiotherapy using deep inspiration breath hold or multi-field intensity modulated radiotherapy, and all non-breast cancer patients will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-08; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To measure the difference in accuracy of a breast imaging protocol that includes a large anterior EPI in detecting set-up errors outside of tolerance as compared to the current standard breast imaging protocols. | Will be measured on days 1, 2 and 3 of radiation therapy and possibly day 4 if adjustments of the EPI where required.

SECONDARY OUTCOMES:
What effect does the addition of a larger anterior EPI have on detection of setup errors in the medial/lateral, anterior/posterior, or superior/inferior directions and at what frequency do these errors occur in clinical practice. | Will be measured on days 1, 2 and 3 of radiation therapy and possibly day 4 if adjustments of the EPI where required.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Wai, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BCCA - Vancouver Island Cancer Centre, Victoria, British Columbia, Canada